CLINICAL TRIAL: NCT03392441
Title: Pilot Study to Evaluate the Effects of Insulin Deprivation on Brain Structure and Function in Humans With Type 1 Diabetes
Brief Title: Insulin Deprivation on Brain Structure and Function in Humans With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, K. Sreekumaran Nair, Consultant Endocrinology and Metabolism, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17-005244
Record Dates: First submitted 2017-12-13; First posted 2018-01-08 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes; Diabetes Complications
Keywords: dementia; cognition; insulin; adolescent
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Diabetes Complications; Dementia; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Insulin Deprivation (Experimental): Insulin Deprivation in Type 1 Diabetic Patients will be performed for a short time period (4-6 hours). Changes to Age, Sex, and Gender matched controls will be compared.
  Interventions: Other: Insulin Deprivation in Type 1 Diabetic Patients

INTERVENTIONS:
Other: Insulin Deprivation in Type 1 Diabetic Patients — Type 1 Diabetic Patients requiring insulin will have insulin stopped for a short period of time (4-6 hours)

SUMMARY:
What are the effects of transient insulin deprivation on brain structure, blood flow, mitochondrial function, and cognitive function in T1DM patients?

What are the effects of transient insulin deprivation on circulating exosomes and metabolites in T1DM patients?

DETAILED DESCRIPTION:
Diabetes is associated with impaired cognition, abnormal brain development in children, and dementia in older adults, however the underlying mechanisms remain unclear. Little is known about the brain-specific effects of acute insulin deficiency. Our recent studies in diabetic mice show an overall down regulation of brain mitochondrial ATP production and up regulation of several key mitochondrial proteins, indicating that insulin withdrawal has a profound effect on brain mitochondria as well as proteins implicated in neurodegeneration. Hyperglycemia is known to alter cognitive function, but it is unclear if insulin deprivation independently alters cognitive function and has not been assessed in humans.

In order to investigate the effects of insulin deprivation on the human brain, we propose a study involving temporary insulin deprivation in adolescents and adults with type 1 diabetes (T1DM). We will perform brain MRI, phosphorus31 spectroscopy, cognitive testing, circulating blood exosome measurements, and proteomics from muscle biopsy; comparing these measures during insulin treatment and deprivation between diabetic patients and age-, sex-, BMI-matched controls.

Specific aim 1: Determine whether transient insulin deprivation in T1DM adults and adolescents alters brain structure, functions and blood flow as assessed by structural/functional MRI.

Specific aim 2: Determine whether transient insulin deprivation in T1DM adults and adolescents alters cognitive function.

Specific aim 3: Determine whether transient insulin deprivation in T1DM adults and adolescents alters the circulating blood exosome contents and metabolome that can potentially impact brain functions.

Specific aim 4: Determine whether transient insulin deprivation in T1DM adults alters the skeletal muscle proteome homeostasis especially those involved in fission and fusion

ELIGIBILITY:
Inclusion criteria:

* Male and females age 14-17 years, females must be post-menarcheal
* Age 18-45 years
* Able to provide written consent
* Parents able to provide written consent
* T1DM treated with CSII or MDI (not degludec)

Exclusion criteria:

* BMI < 20 or > 30 kg/m2
* BMI z-score <5th or >95th percentile
* Celiac disease
* Pregnancy
* Smoking
* Reported history of illicit substance use
* History of active cardiovascular, cerebrovascular, or peripheral vascular disease
* Active renal disease evidenced by estimated GFR < 50 mL/min/1.73 m2
* History of traumatic brain injury
* Dementia or any other neurologic disease
* Psychiatric disease\
* Any learning disability
* Hemoglobin A1c > 8.5%
* Hemoglobin A1c > 9%
* T2DM, or impaired fasting glucose

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2019-07-05 (Actual)

PRIMARY OUTCOMES:
Change in Structural MRI | baseline, 6 hours
  Structural magnetic resonance imaging (MRI) is a non-invasive technique for examining the anatomy and pathology of the brain (as opposed to using functional magnetic resonance imaging [fMRI] to examine brain activity. This produces images which can be used for clinical radiological reporting as well as for detailed analysis.

CONTACTS AND LOCATIONS:
Overall Officials: K Sreekumaran Nair, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Creo AL, Cortes TM, Jo HJ, Huebner AR, Dasari S, Tillema JM, Lteif AN, Klaus KA, Ruegsegger GN, Kudva YC, Petersen RC, Port JD, Nair KS. Brain functions and cognition on transient insulin deprivation in type 1 diabetes. JCI Insight. 2021 Mar 8;6(5):e144014. doi: 10.1172/jci.insight.144014. PMID 33561011
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials